CLINICAL TRIAL: NCT02155166
Title: Effect of Injectable Intracervical Anesthesia on the Pain Associated With the Insertion of the Levonorgestrel-releasing Intrauterine System in Women Without Previous Vaginal Delivery: a Randomized Controlled Trial
Brief Title: Effect of Intracervical on the Pain Associated With the Insertion of the LNG-IUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Carolina Sales Vieira, Medical Doctor, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNG-IUS-2
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Pain
Keywords: Levonorgestrel-releasing intrauterine system; anesthesia; pain; nulliparous
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intracervical anesthesia (Active Comparator): Intracervical anesthesia with lidocaine 2%
  Interventions: Drug: Intracervical anesthesia with lidocaine 2%
- ibuprofen (Active Comparator): ibuprofen 400 mg
  Interventions: Drug: ibuprofen 400 mg

INTERVENTIONS:
Drug: Intracervical anesthesia with lidocaine 2% — 5 min before LNG-IUS placemen
  Arms: intracervical anesthesia
Drug: ibuprofen 400 mg — 1 hour prior to the LNG-IUS insertion
  Arms: ibuprofen

SUMMARY:
This study has the objective to evaluate the effect of Injectable intracervical anesthesia in comparison with a non-steroidal anti-inflammatory drug (NSAID) on the pain scores immediately after insertion of the levonorgestrel-releasing intrauterine system (LNG-IUS) in women without previous vaginal delivery.

H0: There is no difference in terms of pain score between the treatments H1: There will be difference in terms of pain score between treatments

DETAILED DESCRIPTION:
Objective: To evaluate the effect of Injectable intracervical anesthesia in comparison with a non-steroidal anti-inflammatory drug (NSAID) on the pain scores immediately after insertion of the levonorgestrel-releasing intrauterine system (LNG-IUS) in women without previous vaginal delivery. As secondary objectives, the effects of the interventions on the pain scores assessed 2 and 6 hours after the LNG-IUS insertion, the level of discomfort associated with the insertion procedure and the ease of insertion of the LNG-IUS will be evaluated.

Design: open randomized controlled trial Setting: Outpatient contraceptive services Patients: 100 women who want to use the LNG-IUS Interventions: 100 women will be randomized into two groups: a) use of a NSAID (ibuprofen, 400 mg) 1 hour before the LNG-IUS insertion; and b) 2% lidocaine intracervical injection. These women will be evaluated immediately after the LNG-IUS insertion, and then 2 hours and 6 hours after it.

Main outcome measures: Two pain scales will be used (the visual analogue scale and the facial pain scale) in addition to assessing the ease of insertion (as rated by the provider) and the level of discomfort from the procedure (as rated by the patient). Multivariate logistic regression will be performed to analyze the predictors associated with moderate/severe pain.

ELIGIBILITY:
Inclusion Criteria:

* patients who wanted to use the LNG-IUS as a contraceptive
* age between 18 and 45 years
* nulliparity
* absence of previous vaginal delivery

Exclusion Criteria:

* women in categories 3 and/or 4 for LNG-IUS use according to the medical eligibility criteria of the World Health Organization
* illicit drug and/or alcohol users
* women with allergies or contraindications to NSAIDs or lidocaine
* chronic pelvic pain of any etiology
* abnormalities in the cervix (such as fibrosis or isthmus-cervical incompetence)
* previous abortion with or without uterine curettage
* psychiatric disorders
* continued use of medications that could interfere with the pain threshold

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain | immediately after LNG-IUS insertion (approx 1 sec)
  Pain associated with the levonorgestrel-releasing intrauterine system (LNG-IUS) insertion (by visual analogue scale and face scale)

SECONDARY OUTCOMES:
Pain | 2 and 6 hours after the LNG-IUS insertion
  To evaluate the effects of the interventions on the pain scores assessed 2 and 6 hours after the LNG-IUS placement (by by visual analogue scale and face scale)
Discomfort | immediately after LNG-IUS insertion (approx 1 sec)
  To evaluate the level of discomfort associated with the LNG-IUS insertion (By the experience of the patient in terms of LNG-IUS as slightly uncomfortable, uncomfortable, or very uncomfortable)
ease of insertion | immediately after LNG-IUS insertion (approx 1 sec)
  To evaluated the ease of insertion of the LNG-IUS (as rated by the provider)

CONTACTS AND LOCATIONS:
Overall Officials: CAROLINA S VIEIRA, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] Castro TV, Franceschini SA, Poli-Neto O, Ferriani RA, Silva de Sa MF, Vieira CS. Effect of intracervical anesthesia on pain associated with the insertion of the levonorgestrel-releasing intrauterine system in women without previous vaginal delivery: a RCT. Hum Reprod. 2014 Nov;29(11):2439-45. doi: 10.1093/humrep/deu233. Epub 2014 Sep 19. PMID 25240012